CLINICAL TRIAL: NCT06802965
Title: Shanghai Atrial Fibrillation Registry
Acronym: SAFE
Status: Enrolling by invitation | Type: Observational
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Shanghai Health Statistics Center (Unknown)
Responsible Party: Principal Investigator, Yiguang LI, Dr, Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Other Study IDs: XHEC-C-2024-220-1
Record Dates: First submitted 2025-01-26; First posted 2025-01-31 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Atrial Fibrillation (AF)
Keywords: atrial fibrillation; left atrial appendage closure; catheter ablation; risk score; Chinese
MeSH Terms: conditions — Atrial Fibrillation | interventions — Catheter Ablation; Left Atrial Appendage Closure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with AF: All patients with a diagnosis of AF and residents of Shanghai are included.
  Interventions: Procedure: catheter ablation, left atrial appendage closure

INTERVENTIONS:
Procedure: catheter ablation, left atrial appendage closure — Compare the clinical prognosis of patients with AF underwent the combined procedure of catheter ablation and left atrial appendage closure (LAAC), single catheter ablation and single LAAC.

SUMMARY:
Using the Shanghai Municipal Health Commission database and Shanghai Centers for Disease Control and Prevention database, patients with AF in Shanghai are included to construct the Shanghai AF registry to investigate clinical characteristics, treatment, and prognosis.

DETAILED DESCRIPTION:
1. To determine the most suitable risk stratification model for Chinese AF population regarding stroke and major cardiovascular events, i.e. CHA2DS2-VASc, CHA2DS2-VASc-60, or CHA2DS2-VA scores.
2. To compare the clinical prognosis of patients with AF receiving the combined procedure of catheter ablation and left atrial appendage closure (LAAC), single catheter ablation, and single LAAC.

ELIGIBILITY:
Inclusion Criteria:

* With diagnosis of AF: the diagnosis must be identified from the Shanghai Municipal Health Commission database and verified by 12-lead ECG or Holter monitoring since 2015
* Residents of Shanghai
* Taking part in the government-issued health insurance, including the Urban Residents' Basic Medical Insurance (URBMI), the Urban-Employ Based Medical Insurance (UEBMI) and the New Rural Cooperative Medical Scheme (NRCMS).

Exclusion Criteria:

* Non-residence of Shanghai
* Without the government-issued health insurance
* Die at the day of index diagnosis of AF

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population include patients with a diagnosis of AF in the Shanghai Municipal Health Commission database who are residence of Shanghai and with government-issued health insurance.
Sampling Method: Non-Probability Sample
Enrollment: 400000 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
Composite of death, ischemic stroke, systemic embolism, myocardial infarction, major bleeding, and acute heart failure | From enrollment to December 31, 2024
  Composite of death, ischemic stroke, systemic embolism, myocardial infarction, major bleeding, and acute heart failure

SECONDARY OUTCOMES:
Cardiovascular death | From enrollment to December 31, 2024
  Death due to the following reasons: Ischemic heart diseases; Hypertensive heart diseases; Other heart and vascular diseases, including myocarditis, endocarditis, pulmonary embolism, aortic aneurysm, dissecting aneurysm; Sudden, unexpected, and unwitnessed death or death of unknown cause; Ischemic stroke; Hemorrhagic stroke and non-traumatic intracranial bleeding
Non-cardiovascular death | From enrollment to December 31, 2024
  Death caused by: Alzheimer's disease, Parkinson's disease, other neurological diseases except vascular central nervous system causes; Diabetes mellitus; Cancers (malignant solid tumors); Chronic obstructive pulmonary disease, lower respiratory infections, and other respiratory diseases; Gastrointestinal and liver diseases; Chronic kidney diseases and other kidney diseases; Leukemia, lymphoma, and other diseases of blood system; Falls; Road injuries; Drowning and asphyxia; Self-harm; COVID-19; Other non-cardiovascular causes of death, etc.
Ischemic stroke | From enrollment to December 31, 2024
  * Neurological deficit of cerebrovascular cause that persists beyond 24 hours or is interrupted by death within 24 hours.
  * Exclusion of coma due to severe brain trauma, intracranial tumor, metabolic disorder or fluid or electrolyte imbalance, peripheral neuropathy, or CNS infection.
  * Not meeting criteria for subarachnoid hemorrhage, intraparenchymal hemorrhage and other hemorrhage
  * With imaging findings
Systemic embolism | From enrollment to December 31, 2024
  * Acute vascular insufficiency or occlusion of the extremities or any non-CNS organ associated with clinical, imaging, surgical/autopsy evidence of arterial occlusion.
  * Exclusion of other likely mechanism, e.g., trauma, atherosclerosis, or instrumentation, etc.
Myocardial infarction | From enrollment to December 31, 2024
  * A rise of cardiac biomarker values (preferably cardiac troponin) with at least one value above the 99th percentile upper reference limit and with at least one of the following:
  * Symptoms of ischemia
  * ECG evidence: new ST-segment-T wave (ST-T) changes, or new left bundle branch block, or new pathological Q waves
  * Imaging evidence: new loss of viable myocardium or new regional wall motion abnormality
  * Angiography evidence: intracoronary thrombus
Major bleeding | From enrollment to December 31, 2024
  At least one of the following conditions:
  * Fatal bleeding
  * Symptomatic bleeding in a critical organ, such as intracranial, intraspinal, intraocular, retroperitoneal, intra-articular or pericardial, or intramuscular with compartment syndrome
  * Bleeding causing a fall in hemoglobin level of 20 g/L or more or leading to transfusion of two or more units of whole blood or red cells.
Acute Heart failure (HF) | From enrollment to December 31, 2024
  * Hospitalization, or emergency department visit requiring treatment with infusion therapy, for a clinical syndrome that presents with multiple signs and symptoms consistent with cardiac decompensation or inadequate cardiac pump function.
  * Evidence in the doctor's notes that the reason for this hospitalization, or emergency department visit, was heart failure.
  * Evidence of signs and symptoms: increasing or new onset shortness of breath, edema, paroxysmal nocturnal dyspnea, orthopnea, and hypoxia
  * Include acute decompensated HF with preserved, mid-range, and reduced left ventricular ejection fraction.
  * If a patient was diagnosed and treated for HF in an outpatient setting without infusion therapy for decompensated HF, such condition was not considered an outcome.

OTHER OUTCOMES:
Medical cost | From enrollment to December 31, 2024
  Medical cost related to: AF and non-AF diseases; at emergency department, outpatient and inpatient.

CONTACTS AND LOCATIONS:
Locations (1):
- Xinhua Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No